CLINICAL TRIAL: NCT06948825
Title: Effectiveness Study of a Lifestyle Intervention Versus Metformin in Mothers With Recent Gestational Diabetes
Acronym: GooDMomS2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: University of North Carolina (Other); Diabetes Sisters (Unknown); American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 48359-1-ECNS91615N
Record Dates: First submitted 2025-03-26; First posted 2025-04-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Weight Loss; Gestational Diabetes Mellitus in Pregnancy; Postpartum Care
Keywords: diabetes prevention; gestational diabetes; lifestyle intervention
MeSH Terms: conditions — Weight Loss; Diabetes, Gestational | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Adaptive trial design. All participants receive the basic lifestyle intervention. If they do not reach their weight loss threshold, they are then randomized to an enhanced lifestyle intervention or Metformin.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Enhanced Lifestyle (eLI) (Active Comparator): Participants will continue with the same components as the Lifestyle Intervention (LI), with the addition of guidance on healthy meal planning and online grocery shopping, including one free delivery per week via instacart. If randomized to this group, participants will continue to have group sessions every other week with others in the eLI arm of the study for the duration of the study (5 or 4.5 months depending on when they were randomized to the Metformin arm) for a total of a 6-month intervention. Group sessions will last 45-60 minutes each. These sessions will be led by a trained health counselor.
  Interventions: Behavioral: Enhanced Lifestyle Intervention
- Metformin arm (MI) (Active Comparator): Participants in this arm will have an individual in-person session with the health counselor and study provider where they receive information about 1) the risks and benefits of Metformin for weight loss, 2) potential risks of infant hypoglycemia and the signs/symptoms of infant hypoglycemia, 3) risk factors for development of infant hypoglycemia and the potential long-term effects and consequences of infant hypoglycemia and, 4) guidance on how to take Metformin.
  Participants will be placed on Metformin by mouth (850 mg daily x 7 days, then 850 mg twice daily) and will have a 15-minute follow-up call one week after starting the medication to answer additional questions, assess for any medication side effects, and assess for adherence, and then 15-minute follow-up calls by the research team every 2 weeks. Participants will be encouraged to continue practicing healthy lifestyle behaviors learned during the first 4 weeks of the intervention.
  Interventions: Drug: Metformin Hcl 850Mg Tab
- Lifestyle Intervention (LI) (Active Comparator): All participants will begin with the DPP-based Lifestyle Intervention (LI). This arm includes weekly online 45-minute Zoom group sessions for 4 weeks. After week 4, Zoom group sessions will be biweekly. The goal is a 2% weight loss at 4 weeks and a 3% weight loss at 6 weeks. If participants reach their weight loss goal, they will continue in this arm of the study. These sessions will be led by a trained health counselor.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Drug: Metformin Hcl 850Mg Tab — Participants randomized to Metformin will have a prescription of Metformin 850mg orally twice a day. The participant will get blood drawn for testing, undergo a urine pregnancy test, and meet with the study provider to discuss the medication.
  Arms: Metformin arm (MI)
Behavioral: Lifestyle Intervention — Participants in the Lifestyle Intervention will meet once a week via zoom with the study health counselor to go over lesson plans. After 4 weeks, participants will meet via zoom every other week.
  Arms: Lifestyle Intervention (LI)
Behavioral: Enhanced Lifestyle Intervention — Participants in the Enhanced Lifestyle Intervention will meet every other week, and will get a free instacart membership to have access to free grocery delivery. Additionally, participants in this intervention will have a 1:1 virtual meeting focused on meal planning with the study health counselor.
  Arms: Enhanced Lifestyle (eLI)

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a 6-month lifestyle intervention compared to Metformin in postpartum women who have delivered a singleton, live born infant within the last 12 weeks to 1 year and had a pregnancy complicated by gestational diabetes. The main question this study aims to answer is:

Is a Lifestyle Intervention or Metformin more effective for weight loss in postpartum women with recent gestational diabetes?

Researchers will compare a 6-month Lifestyle Intervention and Metformin to see if either intervention is more effective in achieving weight loss and improving health outcomes.

Participants will:

* Attend an in-person baseline visit to receive a Bluetooth-enabled scale and Fitbit, have blood drawn for testing, and have their height, weight, and blood pressure measured. Participants will also be asked to bring in their infant, and the study team will measure the infant's weight and length.
* Track diet, physical activity, and weight using the Fitbit and Looseit! apps.
* Attend weekly online group sessions for the first 4 weeks, then biweekly sessions.
* If not meeting weight loss goals, be randomized to either Enhanced Lifestyle Intervention or Metformin arms of the study.
* If randomized to Metformin, participants will attend one in-person meeting with the study provider, get blood drawn for testing, and undergo a urine pregnancy test before starting the medication.
* Continue with biweekly group sessions or have regular check-in calls.
* If randomized to the Enhanced Lifestyle Intervention, participants will get a free Instacart membership, a 1:1 session with the study health counselor focused on meal planning and free grocery delivery once a week for the remainder of the study.
* Participants will meet every other week via Zoom with the health counselor and other participants in the enhanced lifestyle arm.
* At the end of the 6 months, all participants will come for an in-person visit to get blood drawn for testing. Participants will also be asked to bring in their infant, and the study team will measure the infant's weight and length.

DETAILED DESCRIPTION:
Once enrollment is complete (consent signed), participants will complete the baseline online medical history form and 9 questionnaires available online.

Baseline: Participants will come for an in-person visit to the GW School of Public Health and receive a Bluetooth-enabled digital scale and a Fitbit activity tracker. Research staff will help participants set up a study Fitbit and Looseit! account. Participants will undergo serum blood collection (10 ml) for HgbA1c and lipids. Participants will also be asked to bring in their infant, and the study team will measure the infant's weight and length. Participants will be asked to use this Fitbit and Looseit! account for the duration of the study to track their diet, activity, and weight. Study staff will access this data, review participant progress, and provide feedback as needed.

Start: All participants will begin with the DPP-based Lifestyle Intervention (LI). The program includes weekly online 45-minute Zoom group sessions for 4 weeks. After week 4, Zoom group sessions will be biweekly. The goal is a 2% weight loss at 4 weeks and a 3% weight loss at 6 weeks. These sessions will be led by a trained health counselor who is part of the research team. The health counselor will review the Fitbit Tracker information and provide tips for improving dietary intake and physical activity via email or text messaging based on the participant's preference.

At the end of week 4 and week 6, participants will submit their weight through Bluetooth-enabled scales.

If they have reached their weight loss goal, they will continue with the lifestyle intervention (LI) with online Zoom group sessions held every other week for the remainder of the intervention (for a total of a 6-month intervention).

After 4 or 6 weeks, participants who have not yet reached their weight loss goal (non-responders) will be randomly assigned to one of two intervention groups:

1. DPP-based Enhanced Lifestyle intervention (eLI)

   OR
2. Metformin (850 mg daily x 7 days, then 850 mg twice daily) orally

Enhanced Lifestyle Intervention (eLI): Participants will continue with the same components as the Lifestyle Intervention (LI), with the addition of guidance on healthy meal planning and online grocery shopping, including one free delivery per week. If randomized to this group, participants will continue to have group sessions every other week with others in the eLI arm of the study for the duration of the study (5 or 4.5 months, depending on when they were randomized to the Metformin arm) for a total of a 6-month intervention. Group sessions will last 45-60 minutes each. These sessions will be led by a trained health counselor in the research team. The health counselor will review the Fitbit Tracker and looseit! information and provide tips for improving dietary intake and physical activity via email or text messaging based on the participant's preference.

Metformin Arm: Participants in this arm will have an individual in-person session with the health counselor and study provider where they receive information about 1) the risks and benefits of Metformin for weight loss, 2) potential risks of infant hypoglycemia and the signs/symptoms of infant hypoglycemia, 3) risk factors for development of infant hypoglycemia and the potential long-term effects and consequences of infant hypoglycemia and, 4) guidance on how to take Metformin. After the in-person session, participants will visit the LabCorp facility on the GW Foggy Bottom campus to provide 5 mL of serum for creatinine and liver function testing, as well as undergo a urine pregnancy test. Participants with abnormal liver function tests (ALT outside 4-36 U/L or AST outside 8-33 U/L), eGFR < 60 ml/min, or a positive pregnancy test will be ineligible for Metformin. Once lab results are reviewed, participants will be placed on Metformin by mouth (850 mg daily x 7 days, then 850 mg twice daily). Tablets will be distributed by the Investigational Drug Pharmacy at the George Washington School of Medicine and Health Sciences. This is the current dosage prescribed for weight loss in the clinical setting.

Participants on Metformin will have a 15-minute follow-up call one week after starting the medication to answer additional questions, assess for any medication side effects, and assess for adherence, and then 15-minute follow-up calls by the research team every 2 weeks. Participants will be educated that it is safe to continue to breastfeed while on Metformin, as recommended by the American College of Obstetricians and Gynecologists published recommendations on postpartum care following a pregnancy with GDM. There are no group sessions for this group. Participants will be encouraged to continue practicing healthy lifestyle behaviors learned during the first 4 weeks of the intervention.

End of study: At the end of the study (6 months), participants will complete one questionnaire with updates about their health since their baseline questionnaire and will also complete 9 online questionnaires (same as baseline). Participants will come for an in-person visit where they will be asked to bring their pill container, if they were randomized to the Metformin arm, and provide a 10 ml serum sample for HbA1c, and lipids via LabCorp. Participants will also be asked to bring in their infant, and the study team will measure the infant's weight and length.

ELIGIBILITY:
Inclusion Criteria:

* Mothers between 8 weeks and 12 months postpartum from a pregnancy complicated by GDM will be recruited. The research team will begin recruiting women who are at least 8 weeks postpartum to provide time to describe the study and answer any questions. Mothers who want to participate will be enrolled in the study between 12 weeks and 12 months postpartum.
* BMI of 25 kg/m2 to 45 kg/m2
* Singleton delivery
* Participants must also have a working cell phone, be willing to accept email or text messages attend Zoom calls, and be willing to be potentially randomized to drug therapy with Metformin.

Exclusion Criteria:

* Pregnant or planned pregnancy within the next 6 months.
* Participation in any other weight loss program or taking weight loss medication.
* Normal or underweight BMI (BMI < 24.9 kg/m2)
* Multi-fetal (twins or triplets) gestation
* Women with type 1 or type 2 diabetes, malignancy, other serious co-morbidities (advanced kidney disease, NYHA class 3-4 CHF, advanced COPD), schizophrenia or other major psychiatric disease, and substance abuse or AIDS.
* Women whose infants have significant medical conditions, such as congenital heart disease, renal impairment, or hepatic impairment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Mean weight change at 6 months | 6 months
  Weight in kg.

SECONDARY OUTCOMES:
Change in physical activity | 6 months
  Measured using the Paffenberger Physical Activity Questionnaire, scores are calculated as total weekly energy expenditure in kilocalories per week; higher scores indicate better physical activity levels.
Change in blood pressure | 6 months
  Change in blood pressure, measured in mmHg. A better blood pressure reading is considered below 120/80 mmHg.
Change in A1c | 6 months
  Change in A1c lab value, measured in percentage (%), where a better A1c value is below 5.7%.
Change in lipids | 6 months
  Change in lipids, measured in mg/dL, where a better outcome is total cholesterol below 200mg/dL, HDL above 60 mg/dL, LDL below 100 mg/dL, and triglycerides below 150 mg/dL.
Change in quality of life | 6 months
  Measured using the Short-Form Survey 12, where scores range from 0 to 100. Scores higher than 50 indicate better-than-average health.
Change in depression score | 6 months
  Measured using the Edinburgh Postnatal Depression Scale, with scores ranging from 0 to 30, and lower scores indicating better outcomes. A score of 12 or higher indicates the need to connect with a primary care physician or mental health clinician in the GW School of Medicine or the local community. With the participant's permission, the research staff will facilitate this connection.
Change in diet quality | 6 months
  The research team will review participant diet data via the Ascend platform.
Breastfeeding | 6 months
  A question will be asked at the start and end of the study to determine breastfeeding status.
Adherence to Metformin treatment | 4.5 to 5 months
  Participants will complete a Metformin adherence questionnaire every 2 weeks.
Infant weight | 6 months
  Measured in grams.
Infant length | 6 months
  Measured in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Nicholson, MD, Principal Investigator — The George Washington University
Locations (1):
- Milken Institute School of Public Health - The George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share unidentified results of outcomes, including clinical and behavioral outcomes.
Supporting Information: Study Protocol, CSR
Time Frame: 9 months following close of the study.
Access Criteria: Based on a formal request to the principal investigator.

REFERENCES:
- [Background] Ferrara A. Increasing prevalence of gestational diabetes mellitus: a public health perspective. Diabetes Care. 2007 Jul;30 Suppl 2:S141-6. doi: 10.2337/dc07-s206. No abstract available. PMID 17596462
- [Background] DeSisto CL, Kim SY, Sharma AJ. Prevalence estimates of gestational diabetes mellitus in the United States, Pregnancy Risk Assessment Monitoring System (PRAMS), 2007-2010. Prev Chronic Dis. 2014 Jun 19;11:E104. doi: 10.5888/pcd11.130415. PMID 24945238
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Heida KY, Franx A, van Rijn BB, Eijkemans MJ, Boer JM, Verschuren MW, Oudijk MA, Bots ML, van der Schouw YT. Earlier Age of Onset of Chronic Hypertension and Type 2 Diabetes Mellitus After a Hypertensive Disorder of Pregnancy or Gestational Diabetes Mellitus. Hypertension. 2015 Dec;66(6):1116-22. doi: 10.1161/HYPERTENSIONAHA.115.06005. Epub 2015 Oct 12. PMID 26459420
- [Background] Hedderson M, Ehrlich S, Sridhar S, Darbinian J, Moore S, Ferrara A. Racial/ethnic disparities in the prevalence of gestational diabetes mellitus by BMI. Diabetes Care. 2012 Jul;35(7):1492-8. doi: 10.2337/dc11-2267. Epub 2012 May 22. PMID 22619080
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams D. Type 2 diabetes mellitus after gestational diabetes: a systematic review and meta-analysis. Lancet. 2009 May 23;373(9677):1773-9. doi: 10.1016/S0140-6736(09)60731-5. PMID 19465232
- [Background] Hamman RF, Wing RR, Edelstein SL, Lachin JM, Bray GA, Delahanty L, Hoskin M, Kriska AM, Mayer-Davis EJ, Pi-Sunyer X, Regensteiner J, Venditti B, Wylie-Rosett J. Effect of weight loss with lifestyle intervention on risk of diabetes. Diabetes Care. 2006 Sep;29(9):2102-7. doi: 10.2337/dc06-0560. PMID 16936160
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Elmer PJ, Grimm R Jr, Laing B, Grandits G, Svendsen K, Van Heel N, Betz E, Raines J, Link M, Stamler J, et al. Lifestyle intervention: results of the Treatment of Mild Hypertension Study (TOMHS). Prev Med. 1995 Jul;24(4):378-88. doi: 10.1006/pmed.1995.1062. PMID 7479629
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Whelton PK, Appel LJ, Espeland MA, Applegate WB, Ettinger WH Jr, Kostis JB, Kumanyika S, Lacy CR, Johnson KC, Folmar S, Cutler JA. Sodium reduction and weight loss in the treatment of hypertension in older persons: a randomized controlled trial of nonpharmacologic interventions in the elderly (TONE). TONE Collaborative Research Group. JAMA. 1998 Mar 18;279(11):839-46. doi: 10.1001/jama.279.11.839. PMID 9515998
- [Background] Cassina M, Dona M, Di Gianantonio E, Litta P, Clementi M. First-trimester exposure to metformin and risk of birth defects: a systematic review and meta-analysis. Hum Reprod Update. 2014 Sep-Oct;20(5):656-69. doi: 10.1093/humupd/dmu022. Epub 2014 May 25. PMID 24861556
- [Background] Ali MK, Echouffo-Tcheugui J, Williamson DF. How effective were lifestyle interventions in real-world settings that were modeled on the Diabetes Prevention Program? Health Aff (Millwood). 2012 Jan;31(1):67-75. doi: 10.1377/hlthaff.2011.1009. PMID 22232096
- [Background] Phelan S, Hagobian T, Brannen A, Hatley KE, Schaffner A, Munoz-Christian K, Tate DF. Effect of an Internet-Based Program on Weight Loss for Low-Income Postpartum Women: A Randomized Clinical Trial. JAMA. 2017 Jun 20;317(23):2381-2391. doi: 10.1001/jama.2017.7119. PMID 28632867
- [Background] Castorino K, Jovanovic L. Pregnancy and diabetes management: advances and controversies. Clin Chem. 2011 Feb;57(2):221-30. doi: 10.1373/clinchem.2010.155382. Epub 2010 Dec 9. PMID 21148303
- [Background] Syngelaki A, Nicolaides KH, Balani J, Hyer S, Akolekar R, Kotecha R, Pastides A, Shehata H. Metformin versus Placebo in Obese Pregnant Women without Diabetes Mellitus. N Engl J Med. 2016 Feb 4;374(5):434-43. doi: 10.1056/NEJMoa1509819. PMID 26840133
- [Background] American College of Obstetricians and Gynecologists Committee on Practice Bulletins--Obstetrics. ACOG Practice Bulletin. Clinical management guidelines for obstetrician-gynecologists. Number 30, September 2001 (replaces Technical Bulletin Number 200, December 1994). Gestational diabetes. Obstet Gynecol. 2001 Sep;98(3):525-38. PMID 11547793
- [Background] ACOG Committee Opinion No. 736: Optimizing Postpartum Care. Obstet Gynecol. 2018 May;131(5):e140-e150. doi: 10.1097/AOG.0000000000002633. PMID 29683911
- [Background] ACOG Committee Opinion No. 435: postpartum screening for abnormal glucose tolerance in women who had gestational diabetes mellitus. Obstet Gynecol. 2009 Jun;113(6):1419-1421. doi: 10.1097/AOG.0b013e3181ac06b6. PMID 19461459
- [Background] Nicholson WK, Beckham AJ, Hatley K, Diamond M, Johnson LS, Green SL, Tate D. The Gestational Diabetes Management System (GooDMomS): development, feasibility and lessons learned from a patient-informed, web-based pregnancy and postpartum lifestyle intervention. BMC Pregnancy Childbirth. 2016 Sep 21;16(1):277. doi: 10.1186/s12884-016-1064-z. PMID 27654119
- [Background] Refuerzo JS, Viteri OA, Hutchinson M, Pedroza C, Blackwell SC, Tyson JE, Ramin SM. The effects of metformin on weight loss in women with gestational diabetes: a pilot randomized, placebo-controlled trial. Am J Obstet Gynecol. 2015 Mar;212(3):389.e1-9. doi: 10.1016/j.ajog.2014.12.019. Epub 2014 Dec 16. PMID 25526875
- [Background] Hale TW, Kristensen JH, Hackett LP, Kohan R, Ilett KF. Transfer of metformin into human milk. Diabetologia. 2002 Nov;45(11):1509-14. doi: 10.1007/s00125-002-0939-x. Epub 2002 Sep 25. PMID 12436333
- [Background] Gardiner SJ, Kirkpatrick CM, Begg EJ, Zhang M, Moore MP, Saville DJ. Transfer of metformin into human milk. Clin Pharmacol Ther. 2003 Jan;73(1):71-7. doi: 10.1067/mcp.2003.9. PMID 12545145
- [Background] Briggs GG, Ambrose PJ, Nageotte MP, Padilla G, Wan S. Excretion of metformin into breast milk and the effect on nursing infants. Obstet Gynecol. 2005 Jun;105(6):1437-41. doi: 10.1097/01.AOG.0000163249.65810.5b. PMID 15932841
- See also: ACOG Statement on AMA Support for 12 Months of Postpartum Coverage Under Medicaid — http://www.acog.org/news/news-releases/2019/06/acog-statement-on-ama-support-for-12-months-of-postpartum-coverage-under-medicaid